CLINICAL TRIAL: NCT05170191
Title: Effect of Sleep Deprivation on Sensory Integration of Balance, Fall Risk and Postural Stability
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Other Study IDs: FUI/CTR/2021/8
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Sleep Deprivation
Keywords: sleep deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep deprivation: Participant data will be acquired before and after 24 hours of sleep deprivation.
  Interventions: Behavioral: Sleep Deprivation

INTERVENTIONS:
Behavioral: Sleep Deprivation — The participants will stay awake for 24 hours.

SUMMARY:
Sleepiness caused by sleep deprivation may increase the risk of injuries and damages during physical activity. Individual data so far indicates worsening of postural stability and control with females exhibiting better static postural stability regardless of sleeping conditions in comparison to men. However, the literature is deficient in terms of postural stability conditions with eyes open and eyes closed states, as well as fall risk and sensory integration of balance.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 24
* Healthy young adults from Rawalpindi/Islamabad.
* Both males and females
* Participants should have normal sleep patterns without any signs or symptoms of insomnia or hypersomnia.
* Persons without any sleep disorders.
* Persons without any neurological disease.

Exclusion Criteria:

* Persons with sleep disorders such as hypersomnia, insomnia, parasomnia etc.
* Elderly population.
* Persons with any sort of neurological deficits.
* COVID positive and those with any suspected signs and symptoms of COVID-19.
* Alcoholics
* Pregnant females
* A participant with the history of or active diagnosed conditions of any of the following, which renders individual's performance will be excluded:

  * Neurological.
  * Musculoskeletal.
  * Cardiopulmonary.
  * Any congenital disorder or limb deformities.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults aged 19-24 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Postural Stability Index | 24 hours
  Postural stability Index will be measured via Biodex Balance System. A lower score represents better postural stability.
Fall Risk Score | 24 hours
  Fall Risk Score will be measured via Biodex Balance System. A lower score represents better postural stability.
Clinical Test of Sensory Integration and Balance | 24 hours
  Clinical Test of Sensory Integration and Balance will be measured via Biodex Balance System. A lower score represents better postural stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No